CLINICAL TRIAL: NCT03382418
Title: A Phase 1 Double-Blind, Randomized Clinical Trial to Evaluate the Safety and Immunogenicity of a Recombinant Oligomeric gp145 Clade C Env Protein (gp145 C.6980) in Healthy, HIV-1-Uninfected Adult Participants in the US
Brief Title: Evaluating the Safety and Immunogenicity of an HIV Vaccine (gp145 C.6980) in Healthy, HIV-Uninfected Adults in the United States
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 122; 12030 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: gp145 C.6980 (high dose) (Experimental): Participants will receive 300 mcg of the gp145 C.6980 vaccine admixed with aluminum hydroxide adjuvant at Day 0 and Months 2 and 6.
  Interventions: Biological: gp145 C.6980 Vaccine; Biological: Aluminum Hydroxide Adjuvant
- Group 2: gp145 C.6980 (low dose) (Experimental): Participants will receive 100 mcg of the gp145 C.6980 vaccine admixed with aluminum hydroxide adjuvant at Day 0 and Months 2 and 6.
  Interventions: Biological: gp145 C.6980 Vaccine; Biological: Aluminum Hydroxide Adjuvant
- Group 3: Placebo (Placebo Comparator): Participants will receive placebo at Day 0 and Months 2 and 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: gp145 C.6980 Vaccine — Administered by intramuscular injection in the deltoid.
  Other Names: HIV Env gp145 C.6980; recombinant oligomeric gp145 clade C Env protein
  Arms: Group 1: gp145 C.6980 (high dose); Group 2: gp145 C.6980 (low dose)
Biological: Placebo — Sodium Chloride for Injection, 0.9%; Administered by intramuscular injection in the deltoid.
  Arms: Group 3: Placebo
Biological: Aluminum Hydroxide Adjuvant — Administered by intramuscular injection in the deltoid.
  Other Names: Aluminum Hydroxide Suspension
  Arms: Group 1: gp145 C.6980 (high dose); Group 2: gp145 C.6980 (low dose)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of an HIV vaccine (gp145 C.6980) with aluminum hydroxide adjuvant in healthy, HIV-1-uninfected adults in the United States.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immunogenicity of an HIV vaccine (gp145 C.6980) with aluminum hydroxide adjuvant in healthy, HIV-1-uninfected adults in the United States.

Participants will be randomly assigned to one of three groups. Participants in Group 1 will receive 300 mcg of gp145 C.6980 and aluminum hydroxide adjuvant on Day 0 and Months 2 and 6. Participants in Group 2 will receive 100 mcg of gp145 C.6980 and aluminum hydroxide adjuvant on Day 0 and Months 2 and 6. Participants in Group 3 will receive placebo on Day 0 and Months 2 and 6.

Study visits will occur at Day 0 (study entry), Weeks 1 and 2, and Months 2, 2.5, 6, 6.25, 6.5, 9, and 12. Visits may include physical examinations, blood and urine collection, HIV testing, risk reduction counseling, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study and completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items initially answered incorrectly
* Agrees not to enroll in another study of an investigational research agent before the last scheduled protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit. Low risk guidelines are found on the protocol web page under Study Materials on the HVTN Members' site (https://members.hvtn.org/protocols/hvtn122).

Laboratory Inclusion Values

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine:

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status:

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until after the last required protocol clinic visit. Effective contraception is defined as using the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception, or
  * Any other contraceptive method approved by the HVTN 122 Protocol Safety Review Team (PSRT),
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 122 study
* Pregnant or breastfeeding
* Active duty and reserve US military personnel

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 122 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made by the HVTN 122 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 122 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 122 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before or scheduled and intended to be received within 14 days after the first vaccination (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled and intended to be received within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of prednisone or equivalent at doses less than 60 mg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency

Clinically significant medical conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Bar, Study Chair — University of Pennsylvania; Hong Van Tieu, Study Chair — New York Blood Center
Locations (3):
- United States (3):
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Tieu HV, Karuna S, Huang Y, Sobieszczyk ME, Zheng H, Tomaras GD, Montefiori DC, Shen M, DeRosa S, Cohen K, Isaacs MB, Regenold S, Heptinstall J, Seaton KE, Sawant S, Furch B, Pensiero M, Corey L, Bar KJ; HVTN 122 Study Team. Safety and immunogenicity of a recombinant oligomeric gp145 subtype C Env protein (gp145 C.6980) HIV vaccine candidate in healthy, HIV-1-uninfected adult participants in the US. Vaccine. 2023 Oct 6;41(42):6309-6317. doi: 10.1016/j.vaccine.2023.07.046. Epub 2023 Sep 9. PMID 37679276

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Vaccine: gp145 C.6980 300 mcg, admixed with Aluminum Hydroxide Suspension to be administered as 1 mL IM in the deltoid at Months 0, 2, and 6
- Group 2: Vaccine: gp145 C.6980, 100 mcg, admixed with Aluminum Hydroxide Suspension to be administered as 1 mL IM in the deltoid at Months 0, 2, and 6
- Group 3: Placebo: Placebo for gp145 C.6980 (Sodium Chloride for Injection, 0.9%) to be administered as 1 mL IM in the deltoid at months 0, 2, and 6
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Started | 25 | 15 | 5
Month .5 Immunogenicity Cohort (HIV uninfected at Month 0.5 and specimen available for assays) | 25 | 14 | 5
Month 6.5 Immunogenicity Cohort (HIV uninfected at Month 6.5 and specimen available for assays) | 21 | 13 | 5
Completed | 22 | 12 | 5
Not Completed | 3 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo | Total
Number analyzed (Participants) | 25 | 15 | 5 | 45
Age, Continuous [Median (Full Range); unit: years] | 26 [18 to 48] | 27 [20 to 46] | 25 [19 to 36] | 26 [18 to 48]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0
  18 - 20 years | 4 | 1 | 1 | 6
  21 - 30 years | 14 | 9 | 2 | 25
  31 - 40 years | 4 | 2 | 2 | 8
  41 - 50 years | 3 | 3 | 0 | 6
  Over 50 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 4 | 29
  Male | 10 | 5 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 5
  Not Hispanic or Latino | 22 | 14 | 4 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 3 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 4 | 0 | 12
  White | 8 | 7 | 4 | 19
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 15 | 5 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. Corrected Version 2.1, dated July 2017. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 7 days after first vaccination at Month 0
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Pain and/or Tenderness None | 9 | 4 | 4
  Mild | 14 | 10 | 1
  Moderate | 2 | 1 | 0
  Severe | 0 | 0 | 0
  Life Threatening | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms：Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 7 days after first vaccination at Month 0
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Erythema: None | 25 | 15 | 5
  Erythema: Not Gradable | 0 | 0 | 0
  Erythema: Grade 1: Less than 5 cm diameter | 0 | 0 | 0
  Erythema: Grade 1: Between 6.25 to 25 cm sq area | 0 | 0 | 0
  Erythema: Grade 2: Between 5 to 10 cm diameter | 0 | 0 | 0
  Erythema: Grade 2: Between 25 to 100 cm sq area | 0 | 0 | 0
  Erythema: Grade 3: Greater or equal to 10 cm | 0 | 0 | 0
  Erythema: Grade 3: Greater or equal to 100 cm sq | 0 | 0 | 0
  Erythema: Grade 3: complications | 0 | 0 | 0
  Erythema: Grade 4: complications | 0 | 0 | 0
  Induration: None | 25 | 15 | 5
  Induration: Not Gradable | 0 | 0 | 0
  Induration: Grade 1: Less than 5 cm diameter | 0 | 0 | 0
  Induration: Grade 1: Between 6.25 to 25 cm sq area | 0 | 0 | 0
  Induration: Grade 2: Between 5 to 10 cm diameter | 0 | 0 | 0
  Induration: Grade 2: Between 25 to 100 cm sq area | 0 | 0 | 0
  Induration: Grade 3: Greater or equal to 10 cm | 0 | 0 | 0
  Induration: Grade 3: Greater or equal to 100 cm sq | 0 | 0 | 0
  Induration: Grade 3: complications | 0 | 0 | 0
  Induration: Grade 4: complications | 0 | 0 | 0
  Erythema and/or Induration: None | 25 | 15 | 5
  Erythema and/or Induration: Not Gradable | 0 | 0 | 0
  Erythema and/or Induration: Grade 1: Less than 5 cm diameter | 0 | 0 | 0
  Erythema and/or Induration: Grade 1: Between 6.25 to 25 cm sq area | 0 | 0 | 0
  Erythema and/or Induration: Grade 2: Between 5 to 10 cm diameter | 0 | 0 | 0
  Erythema and/or Induration: Grade 2: Between 25 to 100 cm sq area | 0 | 0 | 0
  Erythema and/or Induration: Grade 3: Greater or equal to 10 cm | 0 | 0 | 0
  Erythema and/or Induration: Grade 3: Greater or equal to 100 cm sq | 0 | 0 | 0
  Erythema and/or Induration: Grade 3: complications | 0 | 0 | 0
  Erythema and/or Induration: Grade 4: complications | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. Corrected Version 2.1, dated July 2017. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Reaction is the maximum of the individual systemic variables for a participant. It does not include temperature.
Time Frame: Measured through 7 days after first vaccination at Month 0
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Malaise and/or fatigue: None | 18 | 9 | 4
  Malaise and/or fatigue: Mild | 5 | 5 | 0
  Malaise and/or fatigue: Moderate | 2 | 1 | 1
  Malaise and/or fatigue: Severe | 0 | 0 | 0
  Malaise and/or fatigue: Life Threatening | 0 | 0 | 0
  Myalgia: None | 23 | 11 | 5
  Myalgia: Mild | 2 | 4 | 0
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Life Threatening | 0 | 0 | 0
  Headache: None | 20 | 13 | 4
  Headache: Mild | 5 | 2 | 1
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Life Threatening | 0 | 0 | 0
  Nausea: None | 25 | 15 | 4
  Nausea: Mild | 0 | 0 | 1
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Life Threatening | 0 | 0 | 0
  Vomiting: None | 25 | 15 | 5
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Life Threatening | 0 | 0 | 0
  Chills: None | 24 | 15 | 5
  Chills: Mild | 1 | 0 | 0
  Chills: Moderate | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0
  Chills: Life Threatening | 0 | 0 | 0
  Arthralgia: None | 24 | 14 | 5
  Arthralgia: Mild | 1 | 1 | 0
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Life Threatening | 0 | 0 | 0
  Max. Systemic Symptoms: None | 17 | 8 | 2
  Max. Systemic Symptoms: Mild | 6 | 6 | 2
  Max. Systemic Symptoms: Moderate | 2 | 1 | 1
  Max. Systemic Symptoms: Severe | 0 | 0 | 0
  Max. Systemic Symptoms: Life Threatening | 0 | 0 | 0
  Temperature: None | 24 | 15 | 5
  Temperature: Mild | 1 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0
  Temperature: Life Threatening | 0 | 0 | 0

4. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Severity Grade
Description: Severity definitions are found in The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017); For participants reporting multiple AEs over the time frame, the maximum severity grade is counted.
Time Frame: Measured through 30 days after first vaccination at Month 0
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Mild | 6 | 1 | 0
  Moderate | 3 | 2 | 0
  Severe | 0 | 0 | 0
  Potentially Life-threatening | 0 | 0 | 0
  No AE Reported | 16 | 12 | 5

5. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: as for outcome 4
Time Frame: Measured through 30 days after first vaccination at Month 0
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Related | 0 | 0 | 0
  Not Related | 9 | 3 | 0
  No AE Reported | 16 | 12 | 5

6. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: Measured as outlined in Version 2.0 (January 2010) of the Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual)
Time Frame: Measured through 30 days after first vaccination at Month 0
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  SAE | 0 | 0 | 0
  Non-SAE | 9 | 3 | 0
  No AE Reported | 16 | 12 | 5

7. Primary Outcome: Chemistry and Hematology Laboratory Measures With Grade 1 or Higher, Through First Vaccination
Description: Laboratory results are summarized by analyte and timepoint. Analytes and timepoint combinations with grade 1 or higher results are shown.
Time Frame: Measured at 2 weeks after first vaccination
Population: The "overall number of participants analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, or they missed the scheduled visit, or they terminated participation in the study prior to the scheduled visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 14 | 5
Participants
  WBC (1000/cubic mm) | 0 | 0 | 0
  Neutrophils (1000/cubic mm) | 0 | 0 | 0
  Hemoglobin (g/dL) | 0 | 0 | 0
  Lymphocytes (1000/cubic mm) | 0 | 0 | 0
  Platelets (1000/cubic mm) | 0 | 0 | 0
  ALT (SGPT) (U/L) | 0 | 0 | 0
  Creatinine (g/dL) | 0 | 0 | 0

8. Primary Outcome: Hematology Laboratory Measures: WBC, Neutrophils , Lymphocytes and Platelets
Description: For each chemistry laboratory measure, summary statistics were presented by analyte and treatment group for the overall population.
Time Frame: Measured at 2 weeks after first vaccination
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 14 | 5
thousand cells/cubic mm
  WBC (1000/cubic mm) | 6.10 [5.27 to 7.12] | 5.95 [4.70 to 7.61] | 6.80 [6.20 to 7.51]
  Neutrophils (1000/cubic mm) | 3.802 [2.788 to 4.361] | 3.523 [2.950 to 4.940] | 4.114 [3.522 to 4.950]
  Lymphocytes (1000/cubic mm) | 1.750 [1.480 to 2.160] | 1.483 [1.359 to 2.119] | 1.780 [1.778 to 2.009]
  Platelets (1000/cubic mm) | 262 [215 to 295] | 245.5 [226 to 300] | 326 [310 to 369]

9. Primary Outcome: Chemistry Laboratory Measures: Hemoglobin, Creatinine
Description: as for outcome 8
Time Frame: Measured at 2 weeks after first vaccination
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 14 | 5
g/dL
  Hemoglobin (g/dL) | 13.50 [12.90 to 14.60] | 12.75 [12.30 to 13.80] | 12.90 [12.00 to 14.20]
  Creatinine (g/dL) | 0.00086 [0.00076 to 0.00090] | 0.00087 [0.00073 to 0.00099] | 0.00076 [0.00075 to 0.00087]

10. Primary Outcome: Chemistry Laboratory Measures: ALT
Description: as for outcome 8
Time Frame: Measured at 2 weeks after first vaccination
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 14 | 5
U/L | 14 [10 to 18] | 15 [12 to 23] | 14 [12 to 15]

11. Secondary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: as for outcome 1
Time Frame: Measured through Month 6.5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  None | 6 | 4 | 4
  Mild | 14 | 10 | 1
  Moderate | 5 | 1 | 0
  Severe | 0 | 0 | 0
  Life Threatening | 0 | 0 | 0

12. Secondary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms：Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through Month 6.5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Erythema and/or Induration: None | 20 | 14 | 4
  Erythema and/or Induration: Not Gradable | 3 | 0 | 1
  Erythema and/or Induration: Grade 1: Less than 5 cm diameter | 0 | 0 | 0
  Erythema and/or Induration: Grade 1: Between 6.25 to 25 cm sq area | 1 | 1 | 0
  Erythema and/or Induration: Grade 2: Between 5 to 10 cm diameter | 0 | 0 | 0
  Erythema and/or Induration: Grade 2: Between 25 to 100 cm sq area | 0 | 0 | 0
  Erythema and/or Induration: Grade 3: Greater or equal to 10 cm | 0 | 0 | 0
  Erythema and/or Induration: Grade 3: Greater or equal to 100 cm sq | 1 | 0 | 0
  Erythema and/or Induration: Grade 3: complications | 0 | 0 | 0
  Erythema and/or Induration: Grade 4: complications | 0 | 0 | 0
  Erythema: None | 20 | 14 | 4
  Erythema: Not Gradable | 4 | 0 | 1
  Erythema: Grade 1: Less than 5 cm diameter | 0 | 0 | 0
  Erythema: Grade 1: Between 6.25 to 25 cm sq area | 1 | 1 | 0
  Erythema: Grade 2: Between 5 to 10 cm diameter | 0 | 0 | 0
  Erythema: Grade 2: Between 25 to 100 cm sq area | 0 | 0 | 0
  Erythema: Grade 3: Greater or equal to 10 cm | 0 | 0 | 0
  Erythema: Grade 3: Greater or equal to 100 cm sq | 0 | 0 | 0
  Erythema: Grade 3: complications | 0 | 0 | 0
  Erythema: Grade 4: complications | 0 | 0 | 0
  Induration: None | 23 | 14 | 5
  Induration: Not Gradable | 0 | 0 | 0
  Induration: Grade 1: Less than 5 cm diameter | 0 | 0 | 0
  Induration: Grade 1: Between 6.25 to 25 cm sq area | 1 | 1 | 0
  Induration: Grade 2: Between 5 to 10 cm diameter | 0 | 0 | 0
  Induration: Grade 2: Between 25 to 100 cm sq area | 0 | 0 | 0
  Induration: Grade 3: Greater or equal to 10 cm | 0 | 0 | 0
  Induration: Grade 3: Greater or equal to 100 cm sq | 1 | 0 | 0
  Induration: Grade 3: complications | 0 | 0 | 0
  Induration: Grade 4: complications | 0 | 0 | 0

13. Secondary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 3
Time Frame: Measured through Month 6.5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Malaise and/or fatigue: None | 14 | 5 | 4
  Malaise and/or fatigue: Mild | 9 | 8 | 0
  Malaise and/or fatigue: Moderate | 2 | 2 | 1
  Malaise and/or fatigue: Severe | 0 | 0 | 0
  Malaise and/or fatigue: Life Threatening | 0 | 0 | 0
  Myalgia: None | 21 | 11 | 4
  Myalgia: Mild | 4 | 4 | 1
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Life Threatening | 0 | 0 | 0
  Headache: None | 16 | 10 | 3
  Headache: Mild | 8 | 5 | 2
  Headache: Moderate | 1 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Life Threatening | 0 | 0 | 0
  Nausea: None | 24 | 13 | 4
  Nausea: Mild | 1 | 1 | 1
  Nausea: Moderate | 0 | 1 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Life Threatening | 0 | 0 | 0
  Vomiting: None | 25 | 15 | 5
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Life Threatening | 0 | 0 | 0
  Chills: None | 23 | 12 | 5
  Chills: Mild | 2 | 3 | 0
  Chills: Moderate | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0
  Chills: Life Threatening | 0 | 0 | 0
  Arthralgia: None | 22 | 14 | 5
  Arthralgia: Mild | 3 | 1 | 0
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Life Threatening | 0 | 0 | 0
  Max. Systemic Symptoms: None | 11 | 5 | 1
  Max. Systemic Symptoms: Mild | 11 | 8 | 3
  Max. Systemic Symptoms: Moderate | 3 | 2 | 1
  Max. Systemic Symptoms: Severe | 0 | 0 | 0
  Max. Systemic Symptoms: Life Threatening | 0 | 0 | 0
  Temperature: None | 24 | 14 | 5
  Temperature: Mild | 1 | 1 | 0
  Temperature: Moderate | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0
  Temperature: Life Threatening | 0 | 0 | 0

14. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: as for outcome 4
Time Frame: Measured through Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Related | 1 | 0 | 0
  Not Related | 14 | 8 | 4
  No AE Reported | 10 | 7 | 1

15. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs), by Severity Grade
Description: as for outcome 4
Time Frame: Measured through Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  Mild | 5 | 4 | 0
  Moderate | 8 | 3 | 4
  Severe | 1 | 1 | 0
  Potentially Life-Threatening | 1 | 0 | 0
  No AE Reported | 10 | 7 | 1

16. Secondary Outcome: Frequency of Serious Adverse Events (SAEs)
Description: as for outcome 6
Time Frame: Measured through Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  SAE | 1 | 0 | 0
  Non-SAE | 14 | 8 | 4
  No Adverse Event Reported | 10 | 7 | 1

17. Secondary Outcome: Chemistry and Hematology Laboratory Results With Grade 1 or Higher, Through All Vaccinations
Description: Laboratory results are summarized by analyte and timepoint. Analytes and timepoint combinations with no grade 1 or higher results are not shown.
Time Frame: Measured during Screening, Month 0.5, 2.5, 6.5 and 9
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: Vaccine: gp145 C.6980 100 mcg, admixed with Aluminum Hydroxide Suspension to be administered as 1 mL IM in the deltoid at Months 0, 2, and 6
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
Participants
  WBC (1000/cubic mm)-Screening | 0 | 0 | 0
  WBC (1000/cubic mm)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  WBC (1000/cubic mm)-Day 14 | 0 | 0 | 0
  WBC (1000/cubic mm)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  WBC (1000/cubic mm)-Day 70 | 0 | 0 | 0
  WBC (1000/cubic mm)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  WBC (1000/cubic mm)-Day 182 | 0 | 0 | 0
  WBC (1000/cubic mm)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  WBC (1000/cubic mm)-Day 273 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)-Screening | 0 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Neutrophils (1000/cubic mm)-Day 14 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Neutrophils (1000/cubic mm)-Day 70 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Neutrophils (1000/cubic mm)-Day 182 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 273: number analyzed (Participants) | 21 | 12 | 4
  Neutrophils (1000/cubic mm)-Day 273 | 0 | 0 | 0
  Hemoglobin (g/dL)-Screening | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Hemoglobin (g/dL)-Day 14 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Hemoglobin (g/dL)-Day 70 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Hemoglobin (g/dL)-Day 182 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  Hemoglobin (g/dL)-Day 273 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)-Screening | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Lymphocytes (1000/cubic mm)-Day 14 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Lymphocytes (1000/cubic mm)-Day 70 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Lymphocytes (1000/cubic mm)-Day 182 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 273: number analyzed (Participants) | 21 | 12 | 4
  Lymphocytes (1000/cubic mm)-Day 273 | 0 | 0 | 0
  Platelets (1000/cubic mm)-Screening | 0 | 0 | 0
  Platelets (1000/cubic mm)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Platelets (1000/cubic mm)-Day 14 | 0 | 0 | 0
  Platelets (1000/cubic mm)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Platelets (1000/cubic mm)-Day 70 | 0 | 0 | 0
  Platelets (1000/cubic mm)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Platelets (1000/cubic mm)-Day 182 | 0 | 0 | 0
  Platelets (1000/cubic mm)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  Platelets (1000/cubic mm)-Day 273 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Screening | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  ALT (SGPT) (U/L)-Day 14 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  ALT (SGPT) (U/L)-Day 70 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 182: number analyzed (Participants) | 21 | 13 | 4
  ALT (SGPT) (U/L)-Day 182 | 0 | 1 | 0
  ALT (SGPT) (U/L)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  ALT (SGPT) (U/L)-Day 273 | 0 | 0 | 0
  Creatinine (g/dL)-Screening | 0 | 0 | 0
  Creatinine (g/dL)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Creatinine (g/dL)-Day 14 | 0 | 0 | 0
  Creatinine (g/dL)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Creatinine (g/dL)-Day 70 | 1 | 0 | 0
  Creatinine (g/dL)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Creatinine (g/dL)-Day 182 | 0 | 0 | 0
  Creatinine (g/dL)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  Creatinine (g/dL)-Day 273 | 1 | 0 | 0

18. Secondary Outcome: Hematology Laboratory Measures: WBC, Platelets, Lymphocytes, Neutrophils , Through All Vaccinations
Description: as for outcome 8
Time Frame: Measured during Screening, Month 0.5, 2.5, 6.5 and 9
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
thousand cells/cubic mm
  WBC (1000/cubic mm)-Screening | 6.20 [5.36 to 7.26] | 6.45 [5.90 to 7.80] | 6.38 [6.30 to 6.50]
  WBC (1000/cubic mm)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  WBC (1000/cubic mm)-Day 14 | 6.10 [5.27 to 7.12] | 5.95 [4.70 to 7.61] | 6.80 [6.20 to 7.51]
  WBC (1000/cubic mm)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  WBC (1000/cubic mm)-Day 70 | 6.00 [5.10 to 7.16] | 7.19 [5.48 to 8.95] | 7.00 [5.30 to 7.10]
  WBC (1000/cubic mm)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  WBC (1000/cubic mm)-Day 182 | 5.90 [5.08 to 6.51] | 7.15 [5.73 to 7.40] | 7.00 [6.45 to 7.55]
  WBC (1000/cubic mm)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  WBC (1000/cubic mm)-Day 273 | 6.75 [5.70 to 8.20] | 6.85 [5.33 to 8.10] | 6.80 [6.55 to 7.65]
  Neutrophils (1000/cubic mm)-Screening | 3.910 [2.797 to 4.699] | 4.180 [3.391 to 4.397] | 3.860 [3.692 to 3.933]
  Neutrophils (1000/cubic mm)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Neutrophils (1000/cubic mm)-Day 14 | 3.802 [2.788 to 4.361] | 3.523 [2.950 to 4.940] | 4.114 [3.522 to 4.950]
  Neutrophils (1000/cubic mm)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Neutrophils (1000/cubic mm)-Day 70 | 3.715 [2.267 to 4.160] | 4.480 [3.191 to 5.372] | 4.040 [3.069 to 4.249]
  Neutrophils (1000/cubic mm)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Neutrophils (1000/cubic mm)-Day 182 | 3.307 [2.440 to 4.178] | 3.930 [3.620 to 5.002] | 3.995 [3.629 to 4.725]
  Neutrophils (1000/cubic mm)-Day 273: number analyzed (Participants) | 21 | 12 | 4
  Neutrophils (1000/cubic mm)-Day 273 | 4.061 [3.117 to 4.849] | 3.998 [2.876 to 4.699] | 4.112 [3.780 to 4.434]
  Lymphocytes (1000/cubic mm)-Screening | 1.670 [1.584 to 2.160] | 1.970 [1.540 to 2.554] | 1.872 [1.790 to 2.048]
  Lymphocytes (1000/cubic mm)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Lymphocytes (1000/cubic mm)-Day 14 | 1.750 [1.480 to 2.160] | 1.483 [1.359 to 2.119] | 1.780 [1.778 to 2.009]
  Lymphocytes (1000/cubic mm)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Lymphocytes (1000/cubic mm)-Day 70 | 1.825 [1.370 to 2.309] | 1.975 [1.627 to 2.407] | 1.888 [1.754 to 2.184]
  Lymphocytes (1000/cubic mm)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Lymphocytes (1000/cubic mm)-Day 182 | 1.818 [1.417 to 2.344] | 1.814 [1.548 to 2.491] | 2.164 [1.871 to 2.434]
  Lymphocytes (1000/cubic mm)-Day 273: number analyzed (Participants) | 21 | 12 | 4
  Lymphocytes (1000/cubic mm)-Day 273 | 2.166 [1.499 to 2.397] | 2.184 [1.636 to 2.704] | 2.014 [1.816 to 2.683]
  Platelets (1000/cubic mm)-Screening | 256.0 [198.0 to 299.0] | 242.0 [219.0 to 322.0] | 334.0 [330.0 to 355.0]
  Platelets (1000/cubic mm)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Platelets (1000/cubic mm)-Day 14 | 262.0 [215.0 to 295.0] | 245.5 [226.0 to 300.0] | 326.0 [310.0 to 369.0]
  Platelets (1000/cubic mm)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Platelets (1000/cubic mm)-Day 70 | 262.0 [207.0 to 330.0] | 239.0 [206.5 to 298.5] | 318.0 [316.0 to 355.0]
  Platelets (1000/cubic mm)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Platelets (1000/cubic mm)-Day 182 | 272.5 [206.0 to 306.0] | 254.0 [219.0 to 308.0] | 342.5 [281.5 to 361.5]
  Platelets (1000/cubic mm)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  Platelets (1000/cubic mm)-Day 273 | 261.5 [211.0 to 314.0] | 250.0 [223.5 to 297.5] | 340.0 [294.5 to 358.5]

19. Secondary Outcome: Chemistry Laboratory Measures: Hemoglobin, Creatinine, Through All Vaccinations
Description: as for outcome 8
Time Frame: Measured during Screening, Month 0.5, 2.5, 6.5 and 9
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
g/dL
  Hemoglobin (g/dL)-Screening | 14.20 [13.40 to 14.80] | 13.60 [13.00 to 14.50] | 14.20 [13.50 to 14.50]
  Hemoglobin (g/dL)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Hemoglobin (g/dL)-Day 14 | 13.50 [12.90 to 14.60] | 12.75 [12.30 to 13.80] | 12.90 [12.00 to 14.20]
  Hemoglobin (g/dL)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Hemoglobin (g/dL)-Day 70 | 13.40 [12.90 to 14.30] | 13.90 [13.05 to 14.75] | 13.30 [12.30 to 14.50]
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Hemoglobin (g/dL)-Day 182 | 13.55 [12.80 to 14.50] | 13.30 [12.40 to 13.80] | 13.40 [12.75 to 14.30]
  Hemoglobin (g/dL)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  Hemoglobin (g/dL)-Day 273 | 13.60 [13.10 to 14.50] | 13.45 [12.75 to 14.05] | 13.80 [12.65 to 14.80]
  Creatinine (g/dL)-Screening | .00082 [.00076 to .00094] | .00084 [.00069 to .00101] | .00078 [.00073 to .00085]
  Creatinine (g/dL)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  Creatinine (g/dL)-Day 14 | .00086 [.00076 to .00090] | .00087 [.00073 to .00099] | .00076 [.00075 to .00087]
  Creatinine (g/dL)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  Creatinine (g/dL)-Day 70 | .00084 [.00075 to .00093] | .00081 [.00078 to .00108] | .00079 [.00076 to .00083]
  Creatinine (g/dL)-Day 182: number analyzed (Participants) | 20 | 13 | 4
  Creatinine (g/dL)-Day 182 | .00086 [.00078 to .00092] | .00079 [.00071 to .00099] | .00083 [.00077 to .00088]
  Creatinine (g/dL)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  Creatinine (g/dL)-Day 273 | .00087 [.00075 to .00096] | .00080 [.00070 to .00096] | .00084 [.00078 to .00092]

20. Secondary Outcome: Chemistry Laboratory Measures: ALT, Through All Vaccinations
Description: as for outcome 8
Time Frame: Measured during Screening, Month 0.5, 2.5, 6.5 and 9
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 15 | 5
U/L
  ALT (SGPT) (U/L)-Screening | 13 [9 to 18] | 14 [12 to 21] | 15 [12 to 16]
  ALT (SGPT) (U/L)-Day 14: number analyzed (Participants) | 25 | 14 | 5
  ALT (SGPT) (U/L)-Day 14 | 14 [10 to 18] | 15 [12 to 23] | 14 [12 to 15]
  ALT (SGPT) (U/L)-Day 70: number analyzed (Participants) | 23 | 12 | 5
  ALT (SGPT) (U/L)-Day 70 | 12 [9 to 18] | 16 [13 to 31] | 12 [12 to 14]
  ALT (SGPT) (U/L)-Day 182: number analyzed (Participants) | 21 | 13 | 4
  ALT (SGPT) (U/L)-Day 182 | 13 [10 to 16] | 15 [13 to 22] | 14 [12 to 20]
  ALT (SGPT) (U/L)-Day 273: number analyzed (Participants) | 22 | 12 | 4
  ALT (SGPT) (U/L)-Day 273 | 13 [11 to 21] | 15 [12 to 24] | 15 [13 to 16]

21. Secondary Outcome: Occurrence of Vaccine-induced Binding Antibodies to HIV Proteins Measured by the Binding Antibody Multiplex Assay (BAMA)
Description: Serum HIV-1-specific IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. Samples from post-enrollment visits have positive responses if they meet three conditions: (1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of pre-vaccination net MFI), (2) net MFI values are greater than 3 times pre-vaccination net MFI, and (3) experimental antigen MFI values are greater than 3 times pre-vaccination MFI. Data are excluded if the blood draw date was outside the allowable window, a participant was HIV-infected, or the reference antigen exceeds 5000 MFI.
Time Frame: Measured at 2 weeks after the first vaccination
Population: "Overall Number of Participants Analyzed" includes those with samples collected at week 2, who were HIV-uninfected and received the first vaccination. "Number Analyzed" counts participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 14 | 5
Participants
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 21 | 13 | 4
  1086C_D7gp120.avi/293F | 0 | 1 | 0
  C.1086C_V1_V2 Tags: number analyzed (Participants) | 21 | 13 | 4
  C.1086C_V1_V2 Tags | 0 | 0 | 0
  Con S gp140 CFI: number analyzed (Participants) | 21 | 13 | 4
  Con S gp140 CFI | 2 | 0 | 0
  gp145 Ref. Std.: number analyzed (Participants) | 21 | 13 | 4
  gp145 Ref. Std. | 1 | 0 | 0
  gp41: number analyzed (Participants) | 21 | 13 | 4
  gp41 | 0 | 0 | 0

22. Secondary Outcome: Level of Vaccine-induced Binding Antibodies to HIV Proteins Measured by the Binding Antibody Multiplex Assay (BAMA)
Description: as for outcome 21
Time Frame: Measured at 2 weeks after the first vaccination
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: mean fluorescent intensity (MFI)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 25 | 14 | 5
mean fluorescent intensity (MFI)
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 21 | 13 | 4
  1086C_D7gp120.avi/293F | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 2.5 [1.0 to 4.8]
  C.1086C_V1_V2 Tags: number analyzed (Participants) | 21 | 13 | 4
  C.1086C_V1_V2 Tags | 1.0 [1.0 to 73.5] | 4.8 [1.0 to 48.0] | 2.0 [1.0 to 4.1]
  Con S gp140 CFI: number analyzed (Participants) | 21 | 13 | 4
  Con S gp140 CFI | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  gp145 Ref. Std.: number analyzed (Participants) | 21 | 13 | 4
  gp145 Ref. Std. | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  gp41: number analyzed (Participants) | 21 | 13 | 4
  gp41 | 357.2 [250.5 to 575.8] | 561.8 [433.8 to 868.2] | 128.5 [92.8 to 547.0]

23. Secondary Outcome: Occurrence of Vaccine-induced Binding Antibodies to HIV Proteins Measured by the Binding Antibody Multiplex Assay (BAMA)
Description: as for outcome 21
Time Frame: Measured at 2 weeks after the third vaccination
Population: "Overall Number of Participants Analyzed" includes those with samples collected at month 6.5, who were HIV-uninfected. "Number Analyzed" counts participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 21 | 13 | 5
Participants
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 17 | 12 | 4
  1086C_D7gp120.avi/293F | 17 | 11 | 0
  C.1086C_V1_V2 Tags: number analyzed (Participants) | 17 | 12 | 4
  C.1086C_V1_V2 Tags | 0 | 0 | 0
  Con S gp140 CFI: number analyzed (Participants) | 17 | 12 | 4
  Con S gp140 CFI | 17 | 12 | 0
  gp145 Ref. Std: number analyzed (Participants) | 17 | 12 | 4
  gp145 Ref. Std | 17 | 12 | 0
  gp41: number analyzed (Participants) | 17 | 12 | 4
  gp41 | 17 | 12 | 0

24. Secondary Outcome: Level of Vaccine-induced Binding Antibodies to HIV Proteins Measured by the Binding Antibody Multiplex Assay (BAMA)
Description: as for outcome 21
Time Frame: Measured at 2 weeks after the third vaccination
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: mean fluorescent intensity (MFI)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 21 | 13 | 5
mean fluorescent intensity (MFI)
  1086C_D7gp120.avi/293: number analyzed (Participants) | 17 | 12 | 4
  1086C_D7gp120.avi/293 | 12189.8 [5289.0 to 23738.8] | 7134.2 [2782.3 to 16839.1] | 1.0 [1.0 to 1.6]
  C.1086C_V1_V2 Tags: number analyzed (Participants) | 17 | 12 | 4
  C.1086C_V1_V2 Tags | 20.2 [2.8 to 84.5] | 20.1 [2.5 to 99.8] | 2.4 [1.0 to 4.5]
  Con S gp140 CFI: number analyzed (Participants) | 17 | 12 | 4
  Con S gp140 CFI | 30999.8 [26800.2 to 32050.8] | 22801.4 [9093.4 to 28761.4] | 1.0 [1.0 to 1.0]
  gp145 Ref. Std: number analyzed (Participants) | 17 | 12 | 4
  gp145 Ref. Std | 30210.0 [27178.0 to 32214.8] | 24435.8 [7701.4 to 29542.5] | 1.0 [1.0 to 1.0]
  gp41: number analyzed (Participants) | 17 | 12 | 4
  gp41 | 30111.0 [24748.2 to 32133.5] | 20853.0 [11732.1 to 29509.4] | 137.8 [76.4 to 475.3]

25. Secondary Outcome: Occurrence of HIV-specific CD4+ and CD8+ T-cell Responses to the HIV Proteins Included in the Vaccine. Measured by Flow Cytometry.
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers after peptide stimulation minus % cells expressing markers after no stimulation. A contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). A one-sided Fisher's exact test is applied, testing if the number of cells positive for the marker is equal in the stimulated vs. unstimulated cells. A discrete Bonferroni adjustment is made over the peptide pools. Response is positive if p<=0.00001. Data are excluded if the blood draw date was outside the visit window, the participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high.
Time Frame: Measured at 2 weeks after the third vaccination
Population: "Overall Number of Participants Analyzed" includes those with samples collected at the month 6.5 immunogenicity timepoint, who were HIV-uninfected. "Number Analyzed" counts participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 20 | 13 | 5
Participants
  CD4+: ANY ENV PTEG | 7 | 5 | 0
  CD4+: ENV-1-PTEG-SEQ | 5 | 3 | 0
  CD4+: ENV-2-PTEG-SEQ | 7 | 5 | 0
  CD4+: ENV-3A-PTEG-SEQ: number analyzed (Participants) | 19 | 13 | 5
  CD4+: ENV-3A-PTEG-SEQ | 0 | 0 | 0
  CD4+: ENV-3B-PTEG-SEQ | 0 | 0 | 0
  CD8+: ANY ENV PTEG | 0 | 0 | 1
  CD8+: ENV-1-PTEG-SEQ | 0 | 0 | 0
  CD8+: ENV-2-PTEG-SEQ | 0 | 0 | 1
  CD8+: ENV-3A-PTEG-SEQ | 0 | 0 | 0
  CD8+: ENV-3B-PTEG-SEQ | 0 | 0 | 0

26. Secondary Outcome: Levels of CD4+ and CD8+ T Cells Responses to the HIV Proteins Included in the Vaccine. Measured by Flow Cytometry.
Description: as for outcome 25
Time Frame: Measured at 2 weeks after the third vaccination
Population: "Overall Number of Participants Analyzed" includes those with samples collected at the month 6.5 immunogenicity timepoint, who were HIV-uninfected. "Number Analyzed" shows the number of participants with available data after filtering for assay-specific quality control criteria.
Measure: Median (Inter-Quartile Range); unit: % of T-cell
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 20 | 13 | 5
% of T-cell
  CD4+: ANY ENV PTEG | .109 [.038 to .186] | .117 [.048 to .127] | .008 [.004 to .010]
  CD4+: ENV-1-PTEG-SEQ | .035 [.005 to .058] | .038 [.007 to .048] | -.002 [-.002 to -.001]
  CD4+: ENV-2-PTEG-SEQ | .041 [.026 to .138] | .050 [.021 to .085] | .001 [0 to .004]
  CD4+: ENV-3A-PTEG-SEQ: number analyzed (Participants) | 19 | 13 | 5
  CD4+: ENV-3A-PTEG-SEQ | .006 [.001 to .020] | .007 [.002 to .009] | .009 [.002 to .009]
  CD4+: ENV-3B-PTEG-SEQ | .001 [-.006 to .012] | .001 [-.002 to .007] | .001 [0 to .004]
  CD8+: ANY ENV PTEG | -.004 [-.008 to .010] | -.005 [-.010 to .001] | .008 [.006 to .012]
  CD8+: ENV-1-PTEG-SEQ | 0 [-.004 to .001] | 0 [-.003 to 0] | 0 [0 to 0]
  CD8+: ENV-2-PTEG-SEQ | -.001 [-.004 to .001] | -.003 [-.006 to .001] | .005 [.001 to .012]
  CD8+: ENV-3A-PTEG-SEQ | -.003 [-.006 to .005] | -.002 [-.004 to .002] | .002 [0 to .003]
  CD8+: ENV-3B-PTEG-SEQ | -.001 [-.005 to .006] | -.001 [-.004 to .003] | 0 [-.003 to 0]

27. Secondary Outcome: Occurrence of Neutralizing Antibody Responses Against HIV-1 Isolates
Description: Assessed by multiplex assay. Response to a virus/isolate in the TZM-bl assay is considered positive if the neutralization titer is above a pre-specified cutoff (one-half the lowest dilution tested). A titer is defined as the serum dilution that reduces relative luminescence units (RLUs) by 50% relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only). The pre-specified cutoff is 10 for TZM-bl cells.
Time Frame: Measured at 2 weeks after the third vaccination
Population: "Overall Number of Participants Analyzed" includes those with samples collected at the month 6.5 immunogenicity timepoint, who were HIV-uninfected. "Number Analyzed" shows the number of participants with available data after filtering for assay-specific quality control criteria. Tier 2 isolates data were collected for a subset of participants (9 for group 1, 5 for Group 2, 1 for Group 3).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 21 | 13 | 4
Participants
  Vaccine Strains - 6980.v0.c22 | 0 | 0 | 0
  Tier 1: MW965.26 | 18 | 8 | 0
  Tier 2: 246-F3_C10_2: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: 246-F3_C10_2 | 0 | 0 | 0
  Tier 2: 25710-2.43: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: 25710-2.43 | 0 | 0 | 0
  Tier 2: BJOX002000.03.2: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: BJOX002000.03.2 | 0 | 0 | 0
  Tier 2: CH119.10: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: CH119.10 | 0 | 0 | 0
  Tier 2: CNE55: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: CNE55 | 0 | 0 | 0
  Tier 2: Ce1176_A3: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: Ce1176_A3 | 0 | 0 | 0
  Tier 2: Ce703010217_B6: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: Ce703010217_B6 | 0 | 0 | 0
  Tier 2: TRO.11: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: TRO.11 | 0 | 0 | 0
  Tier 2: X1632-S2-B10: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: X1632-S2-B10 | 0 | 0 | 0

28. Secondary Outcome: Level of Neutralizing Antibody Responses Against HIV-1 Isolates
Description: Assessed by multiplex assay. Response to a virus/isolate in the TZM-bl assay is considered positive if the neutralization titer is above a pre-specified cutoff (one-half the lowest dilution tested). A titer is defined as the serum dilution that reduces relative luminescence units (RLUs) by 50% relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (cells only). The pre-specified cutoff is 10 for TZM-bl cells. Titers below the limit of detection (<10) were set to 5.
Time Frame: Measured at 2 weeks after the third vaccination
Population: as for outcome 27
Measure: Median (Full Range); unit: Titer
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
Number analyzed (Participants) | 21 | 13 | 4
Titer
  Vaccine Strains - 6980.v0.c22 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 1: MW965.26 | 91 [5 to 269] | 30 [5 to 399] | 10 [10 to 10]
  Tier 2: 246-F3_C10_2: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: 246-F3_C10_2 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 2: 25710-2.43: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: 25710-2.43 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 2: BJOX002000.03.2: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: BJOX002000.03.2 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 2: CH119.10: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: CH119.10 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 2: CNE55: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: CNE55 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 2: Ce1176_A3: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: Ce1176_A3 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 2: Ce703010217_B6: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: Ce703010217_B6 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 2: TRO.11: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: TRO.11 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Tier 2: X1632-S2-B10: number analyzed (Participants) | 9 | 5 | 1
  Tier 2: X1632-S2-B10 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected through the month 12 timepoint. All other AEs were collected through 30 days after each vaccination. All-cause mortality were collected through Month 12.
Description: "Other (Not Including Serious) Adverse Events" report participants who had adverse events (not including serious adverse events). Outcome measure 16 report participants who had serious adverse events (1 had, other 14 participants didn't have for Group 1: Vaccine Arm/Group; The participant who had a serious adverse event also had Other (Not Including Serious) Adverse Events; Thus 15 participants in Group 1: Vaccine Arm/Group had Other (Not Including Serious) Adverse Events).
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 15/25 | 8/15 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=25) | Group 2: Vaccine (N=15) | Group 3: Placebo (N=5)
Any SOC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=25) | Group 2: Vaccine (N=15) | Group 3: Placebo (N=5)
Any SOC (Gastrointestinal disorders) | 6 (8) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Any SOC (General disorders) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Any SOC (Infections and infestations) | 7 (9) | 4 (7) | 2 (2)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Any SOC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Any SOC (Investigations) | 5 (6) | 3 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Any SOC (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Any SOC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Any SOC (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Any SOC (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Any SOC (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Any SOC (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Any SOC (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03382418/Prot_001.pdf
  • Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03382418/SAP_002.pdf
  • Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03382418/ICF_000.pdf